CLINICAL TRIAL: NCT03243292
Title: Ten Year Follow-up of Subjects From 3 Landmark Randomized Controlled Bronchial Thermoplasty (BT) Studies
Brief Title: Bronchial Thermoplasty 10+ Year Study
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 92115848
Record Dates: First submitted 2017-07-20; First posted 2017-08-08 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Asthma
Keywords: Bronchial Thermoplasty; Alair; Registry
MeSH Terms: conditions — Asthma | interventions — Bronchial Thermoplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Treated: Subjects that received Bronchial Thermoplasty in a prior study (AIR, RISA, or AIR2)
  Interventions: Other: Bronchial Thermoplasty
- Control: Subjects that participated in prior study (AIR) or (RISA) but did not receive Bronchial Thermoplasty Treatment. Determine if the Control group of subjects asthma has progressed any different from those subjects treated with BT.
  Interventions: Other: Bronchial Thermoplasty
- Sham: Subjects that participated in the AIR2 study, were blinded and did not receive the treatment. Determine if the Sham group of subjects asthma has progressed any different from those subjects treated with BT.
  Interventions: Other: Bronchial Thermoplasty

INTERVENTIONS:
Other: Bronchial Thermoplasty — patients had radio frequency ablation of the smooth muscle for asthma

SUMMARY:
To confirm the long-term efficacy and safety of Bronchial Thermoplasty (BT) at 10 years follow-up or beyond in subjects previously enrolled in any of the following Boston Scientific-sponsored, controlled pre-approval studies: AIR, RISA and AIR2.

DETAILED DESCRIPTION:
Compare rates of severe asthma exacerbations of subjects during the first and fifth year after BT treatment with the proportion of subjects who experience severe asthma exacerbations during the 12 months period prior to enrollment.

Compare baseline HRCT scans from subjects from the AIR2 study that enroll in BT 10+ study to examine if there are any clinically significant post-treatment respiratory changes following BT defined as bronchiectasis or bronchial stenosis.

ELIGIBILITY:
Inclusion Criteria

* Subjects previously enrolled in AIR, RISA or AIR2
* Subjects who received active BT treatment and had last BT treatment at least 10 years and 6 weeks prior to enrollment
* Control/Sham subjects with at least 10 years of long-term follow-up from index date plus 6 weeks
* Subject is able to read, understand and sign a written Informed Consent to participate in the Study and able to comply with the study requirements

Exclusion Criteria:

* Severe asthma exacerbation or chest infection in the past 4 weeks. Subject entry into this study should be delayed until free from severe asthma exacerbation or chest infection for a minimum of 4 weeks.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects that participated in one one or more of the prior studies (AIR, RISA, or AIR2) will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint: Absence of clinically significant post-treatment respiratory changes from Baseline (pre-Bronchial Thermoplasty) CT. | The BT 10+ study's single visit must occur 10 years after the subject's last BT procedure.
  Following BT, defined as bronchiectasis or bronchial stenosis, as confirmed by Pulmonary Volumetric HRCT scan at the BT 10+study visit in those3 subjects who had baseline Volumetric HRCT scan in the AIR2 study. Baseline and 10+ year HRCTs are to be read by an independent radiologist and also assessed by an independent pulmonologist.
Primary Effectiveness: Endpoints at 10 or more years following the subjects' last BT procedure; Asthma Exacerbations, ER Visits, Hospitalizations, and respiratory Serious Adverse Events. | The BT 10+ study's single visit must occur 10 years after the subject's last BT procedure.
  Durability of the treatment effect by comparing the proportion of subjects who experience severe asthma exacerbations during the first and fifth years after BT treatment with the proportion of subjects who experience severe asthma exacerbations during the 12 month period prior to the BT 10+ study visit.

SECONDARY OUTCOMES:
Severe asthma exacerbation rates exacerbations | One day visit
  evaluated for the 12 month period prior to the BT 10+ study visit and will be compared to the first and fifth years after BT treatment:
Severe asthma exacerbation rates subject | One day visit
  evaluated for the 12 month period prior to the BT 10+ study visit and will be compared to the first and fifth years after BT treatment:
Severe asthma exacerbation rates year | One day visit
  evaluated for the 12 month period prior to the BT 10+ study visit and will be compared to the first and fifth years after BT treatment:
rates of emergency room visits for respiratory adverse events | One day visit
  evaluated for the 12 month period prior to the BT 10+ study visit and will be compared to the first and fifth years after BT treatment:
proportion of subjects with emergency room visits for respiratory adverse events | One day visit
  evaluated for the 12 month period prior to the BT 10+ study visit and will be compared to the first and fifth years after BT treatment:
Rates of hospitalizations for respiratory adverse events | One day visit
  evaluated for the 12 month period prior to the BT 10+ study visit and will be compared to the first and fifth years after BT treatment:
Proportion of subjects with hospitalizations for respiratory adverse events | One day visit
  evaluated for the 12 month period prior to the BT 10+ study visit and will be compared to the first and fifth years after BT treatment:
Rates of Respiratory Serious Adverse Events (SAEs) | One day visit
  evaluated for the 12 month period prior to the BT 10+ study visit and will be compared to the first and fifth years after BT treatment:
Proportion of subjects with respiratory SAEs) | One day visit
  evaluated for the 12 month period prior to the BT 10+ study visit and will be compared to the first and fifth years after BT treatment:

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bowman, MD, Study Director — Medical Director, Boston Scientific
Locations (17):
- United States (6):
  - University of Southern California, Los Angeles, California
  - Henry Ford Health System, Detroit, Michigan
  - Regions Hospital Health Partners Specialty Center, Saint Paul, Minnesota
  - Washington University Medical Center, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - Pulmonary Associates of Northern Virginia, Arlington, Virginia
- Brazil (4):
  - Imandade Santa Casa de Misercordia, Pôrto Alegre, Rio Grande do Sul
  - Faculdade da Medicina do ABC, Santo André, São Paulo
  - Gente Clube de Vida Promoção E Serviços 9 Centro de Pesquisa Maimônides, Pôrto Alegre
  - Instituto de Doenças do Tórax /Universidade Federal do Rio de Janeiro/UFRJ, Rio de Janeiro
- Canada (2):
  - Montreal Chest Institute, Montreal, Quebec
  - Institute Universitaire de Cardiologie et Pneumologie de Quebec, Québec, Quebec
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- United Kingdom (4):
  - Chelsea and Westminster Hospital, Chelsea, London
  - Gartnavel General Hospital, Glasgow, Scotland
  - University of Leicester Glenfield Hospital, Leicester
  - Wythenshawe Hospital, University of Manchester, Manchester

REFERENCES:
- [Derived] Chaudhuri R, Rubin A, Sumino K, Lapa E Silva JR, Niven R, Siddiqui S, Klooster K, McEvoy C, Shah PL, Simoff M, Khatri S, Barbers R, Mark Grubb G, McMullen EA, Olson JL, Laviolette M; BT10+ Study Group. Safety and effectiveness of bronchial thermoplasty after 10 years in patients with persistent asthma (BT10+): a follow-up of three randomised controlled trials. Lancet Respir Med. 2021 May;9(5):457-466. doi: 10.1016/S2213-2600(20)30408-2. Epub 2021 Jan 29. PMID 33524320

DOCUMENTS (1):
  • Study Protocol (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT03243292/Prot_000.pdf